CLINICAL TRIAL: NCT01679977
Title: Vibrational-proprioceptive Resistance Exercise Training Versus Neuromuscular Electrical Stimulation Training in Elderly People With Muscle Weakness
Acronym: MOBIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig Boltzmann Institute of Electrical Stimulation and Physical Rehabilitation (Other)
Collaborators: European Union (Other); Ministry of Science and Research, Austria (Unknown); Medical University of Vienna (Other); Comenius University (Other)
Responsible Party: Principal Investigator, Helmut Kern, MD PhD, MD, PhD, Ludwig Boltzmann Institute of Electrical Stimulation and Physical Rehabilitation
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MOBIL
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Muscle Weakness Condition; Therapy Effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Legpress (Active Comparator): Subjects in the LP group train on a custom built, computer controlled, linear electric motor powered leg press device. The so called "swinging" vibrational-proprioceptive mode is used, which means that constant velocity of the pedals (0.3 m/s and 0.2 m/s for concentric and eccentric phase, respectively) are interrupted by short stops (every 8 mm), resulting in short force peaks appearing throughout the movement. Training load is progressively increased throughout the training.
  Interventions: Device: Vibrational-proprioceptive Resistance Exercise Training
- E-Stim (Active Comparator): ES training is performed with a custom-built battery-powered stimulator. The subject are seated over the edge of the therapeutic table with the trunk upright and lower legs freely swinging. Two conductive rubber electrodes covered by wet sponge are placed on the anterior thigh on each side of the body. The electrode pairs are connected to the independent channels of the stimulator and the left and the right thigh are stimulated in an alternative manner. Each repetition (i.e. ES evoked muscle contraction) is evoked by a 3.5 s train (60 Hz) of electrical pulses (rectangular, biphasic, width 0.6 ms). Consecutive contractions of the same thigh are separated by 4.5 s off intervals. Maximal tolerable intensity should be used and is monitored during the training sessions. In all the subjects this should induce a tetanic contraction of the stimulated muscles.
  Interventions: Device: Neuromuscular Electrical Stimulation Training
- Control (No Intervention): This group only perform the same measurements as the intervention groups and lives their live as usual in between.

INTERVENTIONS:
Device: Vibrational-proprioceptive Resistance Exercise Training
  Arms: Legpress
Device: Neuromuscular Electrical Stimulation Training
  Arms: E-Stim

SUMMARY:
Study the structural behaviours of weak muscle of elderly and evaluate the efficiency of two different types of training.

ELIGIBILITY:
Inclusion Criteria:

* age related muscle weakness
* age between 65-85 years
* all inclusion criterias must be fullfilled

Exclusion Criteria:

* recent hip or knee endp-prosthesis (within last 2 years), longstanding immobility
* body mass index greater than 40
* acute thrombosis in lower extremity (within last 3 weeks)
* severe articular effusion
* acute infection
* known myopathy
* relevant neurological diseases with gait disorders (e.g. poly neuropathy, Parkinson's disease)
* dementia, impaired cognitive abilities
* diseases of the vestibular system causing vertigo or impairing balance
* symptomatic cardio pulmonal diseases within the last 6 months
* not or insufficient treated hypertonia
* rheumatic diseases
* other relevant functional impairment of the musculo-skeletal system caused by surgery, trauma or degenerative diseases
* pain in the lower extremity (VAS > 5)
* if one of the above criteria applies the subject will be excluded from the study

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-06; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Maximum voluntary knee extension torque | pre Training, post Training, 3 months post training

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Kern, MD PhD, Study Chair — Ludwig Boltzmann Institute of Electrical Stimulation and Physical Rehabilitation
Locations (2):
- Ludwig Boltzmann Institute of Electrical Stimulation and Physical Rehabilitation, Vienna, Austria
- Facultiy of Physical Education and Sports, Comenius University of Bratislava, Bratislava, Slovakia

REFERENCES:
- [Background] Kern H, Pelosi L, Coletto L, Musaro A, Sandri M, Vogelauer M, Trimmel L, Cvecka J, Hamar D, Kovarik J, Lofler S, Sarabon N, Protasi F, Adami N, Biral D, Zampieri S, Carraro U. Atrophy/hypertrophy cell signaling in muscles of young athletes trained with vibrational-proprioceptive stimulation. Neurol Res. 2011 Dec;33(10):998-1009. doi: 10.1179/016164110X12767786356633. PMID 22196751
- [Background] Sarabon N, Zacirkovnik T, Rosker J, Loefler S. Metric Characteristics of the Tests for Dynamic Balance Evaluation. Phys Med Rehab Kuror. 23(03):135-46, 2013.
- [Background] Sarabon N, Rosker J, Fruhmann H, Burggraf S, Loefler S, Kern H. Reliability of maximal voluntary contraction related parameters measured by a portable isometric knee dynamometer. Phys Med Rehab Kuror. 23(01):22-27, 2013.
- [Background] Mosole S, Rossini K, Kern H, Lofler S, Fruhmann H, Vogelauer M, Burggraf S, Grim-Stieger M, Cvecka J, Hamar D, Sedliak M, Sarabon N, Pond A, Biral D, Carraro U, Zampieri S. Reinnervation of Vastus lateralis is increased significantly in seniors (70-years old) with a lifelong history of high-level exercise (2013, revisited here in 2022). Eur J Transl Myol. 2022 Feb 28;32(1):10420. doi: 10.4081/ejtm.2022.10420. PMID 35234026
- [Background] Vargas Luna JL, Krenn M, Lofler S, Kern H, Cortes R JA, Mayr W. Comparison of Twitch Responses During Current- or Voltage-Controlled Transcutaneous Neuromuscular Electrical Stimulation. Artif Organs. 2015 Oct;39(10):868-75. doi: 10.1111/aor.12623. PMID 26471138
- [Result] Krenn M, Haller M, Bijak M, Unger E, Hofer C, Kern H, Mayr W. Safe neuromuscular electrical stimulator designed for the elderly. Artif Organs. 2011 Mar;35(3):253-6. doi: 10.1111/j.1525-1594.2011.01217.x. PMID 21401669
- [Result] Nejc S, Jernej R, Loefler S, Kern H. Sensitivity of body sway parameters during quiet standing to manipulation of support surface size. J Sports Sci Med. 2010 Sep 1;9(3):431-8. eCollection 2010. PMID 24149637
- [Result] Kern H, Loefler S, Hofer C, Vogelauer M, Burggraf S, Grim-Stieger M, Cvecka J, Hamar D, Sarabon N, Protasi F, Musarò A, Sandri M, Rossini K, Carraro U, Zampieri S. FES Training in Aging: interim results show statistically significant improvements in mobility and muscle fiber size. European Journal Translational Myology - Basic Applied Myology 22(1&2):61-67, 2012.
- [Result] Sarabon N, Rosker J, Loefler S, Kern H. The effect of vision elimination during quiet stance tasks with different feet positions. Gait Posture. 2013 Sep;38(4):708-11. doi: 10.1016/j.gaitpost.2013.03.005. Epub 2013 Apr 6. PMID 23566634
- [Result] Sarabon N, Loefler S, Cvecka J, Sedliak M, Kern H. Strength training in elderly people improves static balance: a randomized controlled trial. European Journal of Translational Myology - Basic Applied Myology 23(3):85-89, 2013.
- [Result] Sedliak M, Cvecka J, Tirpakova V, Loefler S, Sarabon S, Kern H, Hamar D. Reliability of novel postural sway task test. European Journal of Translational Myology - Basic Applied Myology 23(3):81-84, 2013.
- [Result] Kern H, Loefler S, Burggraf S, Fruhmann H, Cvecka J, Sedliak M, Barberi L, De Rossi M, Musarò A, Carraro U, Mosole S, Zampieri S. Elektrostimulation verhindert die Altersbedingte Atrophie der Muskulatur beim Menschen. Eur J of Trans Myol 23(3):105-108, 2013.
- [Result] Hendling M, Krenn M, Haller MA, Loefler S, Kern H, Mayr W. Compliance monitoring of home based electrical stimulation training of elderly subjects. Biomed Tech (Berl). 2013 Aug;58 Suppl 1:/j/bmte.2013.58.issue-s1-A/bmt-2013-4006/bmt-2013-4006.xml. doi: 10.1515/bmt-2013-4006. Epub 2013 Sep 7. No abstract available. PMID 24042616
- [Result] Zampieri S, Pietrangelo L, Loefler S, Fruhmann H, Vogelauer M, Burggraf S, Pond A, Grim-Stieger M, Cvecka J, Sedliak M, Tirpakova V, Mayr W, Sarabon N, Rossini K, Barberi L, De Rossi M, Romanello V, Boncompagni S, Musaro A, Sandri M, Protasi F, Carraro U, Kern H. Lifelong physical exercise delays age-associated skeletal muscle decline. J Gerontol A Biol Sci Med Sci. 2015 Feb;70(2):163-73. doi: 10.1093/gerona/glu006. Epub 2014 Feb 18. PMID 24550352
- [Result] Mosole S, Carraro U, Kern H, Loefler S, Fruhmann H, Vogelauer M, Burggraf S, Mayr W, Krenn M, Paternostro-Sluga T, Hamar D, Cvecka J, Sedliak M, Tirpakova V, Sarabon N, Musaro A, Sandri M, Protasi F, Nori A, Pond A, Zampieri S. Long-term high-level exercise promotes muscle reinnervation with age. J Neuropathol Exp Neurol. 2014 Apr;73(4):284-94. doi: 10.1097/NEN.0000000000000032. PMID 24607961
- [Result] Kern H, Barberi L, Lofler S, Sbardella S, Burggraf S, Fruhmann H, Carraro U, Mosole S, Sarabon N, Vogelauer M, Mayr W, Krenn M, Cvecka J, Romanello V, Pietrangelo L, Protasi F, Sandri M, Zampieri S, Musaro A. Electrical stimulation counteracts muscle decline in seniors. Front Aging Neurosci. 2014 Jul 24;6:189. doi: 10.3389/fnagi.2014.00189. eCollection 2014. PMID 25104935
- [Result] Cvecka J, Tirpakova V, Sedliak M, Kern H, Mayr W, Hamar D. Physical Activity in Elderly. Eur J Transl Myol. 2015 Aug 25;25(4):249-52. doi: 10.4081/ejtm.2015.5280. eCollection 2015 Aug 24. PMID 26913164
- [Result] Zampieri S, Mosole S, Lofler S, Fruhmann H, Burggraf S, Cvecka J, Hamar D, Sedliak M, Tirptakova V, Sarabon N, Mayr W, Kern H. Physical Exercise in Aging: Nine Weeks of Leg Press or Electrical Stimulation Training in 70 Years Old Sedentary Elderly People. Eur J Transl Myol. 2015 Aug 25;25(4):237-42. doi: 10.4081/ejtm.2015.5374. eCollection 2015 Aug 24. PMID 26913162
- [Derived] Mosole S, Carraro U, Kern H, Loefler S, Zampieri S. Use it or Lose It: Tonic Activity of Slow Motoneurons Promotes Their Survival and Preferentially Increases Slow Fiber-Type Groupings in Muscles of Old Lifelong Recreational Sportsmen. Eur J Transl Myol. 2016 Nov 25;26(4):5972. doi: 10.4081/ejtm.2016.5972. eCollection 2016 Sep 15. PMID 28078066